CLINICAL TRIAL: NCT00002288
Title: Safety and Efficacy of Retrovir in HIV Infected Patients Having Neuropsychological Impairments
Brief Title: The Safety and Effectiveness of Retrovir in HIV-Infected Patients Who Have Problems Related to the Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014K; 23
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Neuropsychological Tests; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To assess the efficacy of Retrovir (AZT) therapy in the treatment of HIV Ab positive persons with impairments in neuropsychological functioning. To assess the safety, virologic, and immunologic effects of AZT therapy in HIV Ab positive persons with neuropsychological impairment but minimal other symptomatology.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Neuropsychological (NP) impairments more severe than described in the Inclusion Criteria.
* Evidence of nervous system dysfunction being caused by factors other than HIV infection, including history of head trauma, multiple sclerosis, epilepsy, or presence of concurrent central nervous system (CNS) infections or neoplasms, e.g., toxoplasmosis, primary or metastatic CNS lymphoma, progressive multifocal leukoencephalopathy, cryptococcal or other fungal meningitis, and CNS tuberculous infections.
* Lymphoma or other tumor requiring cytotoxic chemotherapy.

Concurrent Medication:

Excluded:

* Other antiretroviral agents.

Patients with the following are excluded:

* AIDS or advanced ARC.
* Neuropsychological (NP) impairments more severe than described above; i.e., defective performance on NP test battery in 3 or more NP areas on the NP screening battery at 2 standard deviations below the mean.
* Evidence of nervous system dysfunction being caused by factors other than HIV infection, including history of head trauma, multiple sclerosis, epilepsy, or presence of concurrent central nervous system (CNS) metastatic CNS lymphoma, progressive multifocal leukoencephalopathy, cryptococcal or other fungal meningitis, and CNS tuberculous infections.

Prior Medication:

Excluded:

* Antiretroviral agents including zidovudine (AZT).

Prior Treatment:

Excluded within 3 months of study entry:

* Blood transfusion.

Impaired performance on a defined neuropsychological test battery.

* Asymptomatic HIV infection.
* Persistent generalized lymphadenopathy (PGL).
* Early AIDS related complex (ARC).
* Seropositive for human immunodeficiency virus (HIV) demonstrated by positive ELISA test and confirmed by Western blot with no or minimal symptomatology or HIV infection.
* Ability to give informed consent or a person with durable power of attorney who can give informed consent.
* Willingness to be followed by the originating medical center for 1 year.

History of drug or alcohol abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States